CLINICAL TRIAL: NCT06292494
Title: Focused Ultrasound for Drug-resistant Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: InSightec (Industry)
Responsible Party: Principal Investigator, VGHuser_Cheng-Chia Lee, Principal Investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1129052082
Record Dates: First submitted 2023-12-10; First posted 2024-03-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Focused Ultrasound; MR-guided FUS; Drug Refractory Epilepsy; Drug Resistant Epilepsy; Medication Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FUS-treated epilepsy (Experimental)
  Interventions: Device: Exablate 4000 Transcranial MRgfUS System

INTERVENTIONS:
Device: Exablate 4000 Transcranial MRgfUS System — Focused ultrasound interrupt structure of epilepsy network to improve seizure.

SUMMARY:
Focused ultrasound (FUS) has been shown to differentially lesion or modulate (excite and inhibit) brain circuit and neural activity across a broad range of acoustic stimulus parameters (intensity, duty cycle, pulse repetition frequency and pulse duration) for decades. From our previous study, FUS sonication may suppress the number of epileptic signal bursts observed in EEG recordings after the induction of acute epilepsy. The presence of the suppressive effect was found in terms of the number of epileptic EEG spikes from the analysis of the unfiltered and theta-band EEG activity, and further discontinue the seizure attacks. EEG activity has also been consistently reported to have a positive correlation with the level of epilepsy, and FUS-mediated reduction of epileptic EEG activity was most notably observed, no matter lesioning or modulating effects. The aims of this study are to demonstrate the safety and efficacy of FUS technology in epilepsy patients and to estimate the optimal parameters of focused ultrasound exposure that will be used in the case of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 and above.
* Localized refractory epilepsy (ineffective with maximum doses of two or more anti-seizure medications).
* Seizure frequency records for at least one month prior to the trial.
* Patients who have undergone a complete preoperative examination, including EEG, MRI, and positron emission tomography (PET).
* Capable of undergoing high-resolution computed tomography (CT scan), and SDR (Skull Density Ratio) ≥ 0.3.
* Must have a body type suitable for entry into the magnetic resonance imaging (MRI) machine and be able to tolerate MRI scans.
* During the surgical procedure, communication with the physician and the expression of sensory perceptions are essential; general anesthesia is not required.
* Must be able to voluntarily press the stop button.
* Willing to undergo removal of hair from the treatment site.

Exclusion Criteria:

* This product is not suitable for individuals with contraindications related to MRI, such as those with metallic implants, those unable to undergo MRI, severe claustrophobia, or those with adverse reactions to contrast agents.
* Individuals with implants in the brain or skull, such as shunts, electrodes, hard brain membrane patches, or electrode plates, that cannot be avoided along the expected path of brain ultrasound.
* Patients along the expected path of brain ultrasound who cannot avoid structures or sensitive tissues with energy absorption (e.g., previous brain shunt surgery sites, surgical metal clips, or any hard implants).
* Patients with extensive scabbing along the expected path of brain ultrasound.
* Patients who have used contrast agents (e.g., MRI, ultrasound) within the past 24 hours before treatment.
* Patients with other high-risk brain disorders (e.g., intracranial aneurysm).
* Patients with intraoperative or postoperative bleeding risk:

  1. Those with a history of cerebrovascular disease (multiple strokes or strokes within the past six months) or a history of cerebral hemorrhage and stroke.
  2. Those with abnormal bleeding, intracranial bleeding, coagulation disorders, or a history of bleeding or clotting disorders, either during or after surgery.
* Patients taking or injecting anticoagulant medications such as aspirin, coumadin, heparin, novel oral anticoagulants (NOACs), etc., which may lead to prolonged bleeding. Medication should be discontinued for 3-7 days before treatment.
* Patients with severe uncontrolled hypertension (systolic blood pressure > 180 mmHg after stable medication, diastolic blood pressure > 100 mmHg).
* Patients unable to communicate with the physician during the treatment process.
* Unstable cardiac conditions (heart rate > 180 beats/minute or < 40 beats/minute; systolic blood pressure > 180 mmHg or < 90 mmHg).
* Substance abuse (use of illegal drugs or using medications in a manner not recommended by a physician or manufacturer) or alcohol addiction.
* Patients who have taken medications affecting the central nervous system within the past six months (e.g., central nervous system stimulants, sympathomimetic agents).
* Patients with psychological abnormalities (e.g., schizophrenia, severe depression, bipolar disorder).
* Individuals with severe head surface injuries or potential allergies to materials in contact with the head (such as conductive gels, head silicone membranes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pulse rate [Safety] | pre- and post- treatment immediately
  vital sign
blood oxygen saturation level [Safety] | pre- and post- treatment immediately
  vital sign
MRI [Safety] | pre- and post- treatment immediately
  Safety and Tolerability
Incidence of Treatment-Emergent Adverse Events [Tolerability] | during and post- treatment immediately
  To record the adverse events

SECONDARY OUTCOMES:
seizure frequency [efficacy] | pre- and post- treatment immediately and 1,3,6,12 month
  The treatment response is assessed based on the overall observation of seizure frequency.
scalp EEG [efficacy] | pre- and post- treatment immediately and 1,3,6,12 month
  The treatment response is assessed based on the scalp EEG (electroencephalogram).
No. of seizure-free days [efficacy] | pre- and post- treatment immediately and 1,3,6,12 month
  The treatment response is assessed based on the number of seizure-free days within the entire monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chia Lee, MD. PhD., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No